CLINICAL TRIAL: NCT06581042
Title: Understanding Local TReatment Patterns and Outcomes With upAdacitinib in IBD Patients in Belgium
Brief Title: Study to Assess Treatment Patterns and Outcomes With Upadacitinib in Adult Participants With Inflammatory Bowel Disease in Belgium
Status: Recruiting | Type: Observational
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: P24-960
Record Dates: First submitted 2024-08-29; First posted 2024-08-30 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-03

CONDITIONS: Ulcerative Colitis; Crohn's Disease
Keywords: Ulcerative colitis; Crohn's disease; Upadacitinib; RINVOQ
MeSH Terms: conditions — Colitis, Ulcerative; Crohn Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Upadacitinib: Participants will receive upadacitinib as prescribed by their physician according to local label.

SUMMARY:
Crohn's disease (CD) is an incurable chronic inflammatory disorder of the gastrointestinal tract. Ulcerative colitis (UC) is an idiopathic, chronic, inflammatory disease affecting the colon. This study will assess the (long-term) effectiveness and safety of upadacitinib in real-world clinical practice in adult participants with moderate to severe ulcerative colitis (UC) and crohn's disease (CD).

Upadacitinib is an approved drug for treating ulcerative colitis (UC) and Crohn's disease (CD). Approximately 280 participants who are prescribed Upadacitinib by their physician in accordance with local label will be enrolled in 8 sites across Belgium.

Participants will receive upadacitinib as prescribed by their physician according to their routine clinical practice and local label. Participants will be followed for up to 3 years.

There is expected to be no additional burden for participants in this trial. Participants will attend regular visits during the study at a hospital or clinic according to their routine clinical practice

ELIGIBILITY:
Inclusion Criteria:

* Participants with a diagnosis of moderate to severe Crohn's disease or Ulcerative colitis, initiated with upadacitinib at least 12 months prior to inclusion, including participants that were initiated on upadacitinib, but later (i.e. at the moment of data collection) discontinued, or switched to another treatment.
* Participants initiating commercially available upadacitinib at the clinician's discretion as part of their routine clinical care; the decision to administer upadacitinib must be made prior to and independent of recruitment into the study
* Participants prescribed upadacitinib in accordance with the approved local label and treatment recommendations

Exclusion Criteria:

* Participants previously exposed to upadacitinib in a clinical trial or early access program
* Participants participating in interventional research (not including non-interventional
* Participants with stoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult participants with ulcerative colitis or Crohn's Disease
Sampling Method: Non-Probability Sample
Enrollment: 280 (Estimated)
Dates: Start 2024-09-27 (Actual); Primary Completion 2029-09 (Estimated); Study Completion 2029-09 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants Achieving Clinical Remission as per Partial Adapted Mayo Subscores for Ulcerative Colitis | Up to approximately 52 weeks
  Clinical remission is defined as: stool frequency (SF) score < = 1 and not greater than baseline and Rectal bleeding (RB) score = 0
Percentage of Participants Achieving Clinical Remission as per Patient Reported Outcome (PRO2) for Crohn's Disease | Up to approximately 52 weeks
  Clinical remission is defined as stool frequency (SF) score < =3 and not worse than baseline and Abdominal Pain (AP) score < =1 and not worse than baseline

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (7):
- Belgium (7):
  - Imelda Ziekenhuis /ID# 268631, Bonheiden, Antwerpen
  - Universite Libre de Bruxelles - Hopital Erasme /ID# 268632, Anderlecht, Brussels Capital
  - CHU de Liège /ID# 267209, Liège, Liege
  - UZ Gent /ID# 268630, Ghent, Oost-Vlaanderen
  - Vitaz /Id# 268637, Sint-Niklaas, Oost-Vlaanderen
  - AZ Groeninge /ID# 268638, Kortrijk, West-Vlaanderen
  - Groupe Sante CHC - Clinique du MontLegia /ID# 268662, Liège

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=P24-960